CLINICAL TRIAL: NCT06668701
Title: Evaluation of the Naturalistic User Experience of the Website "ich Bin Alles" - an Information Platform for Children and Adolescents with and Without Depression and Their Relatives
Brief Title: Evaluation of the Naturalistic User Experience of the Website "ich Bin Alles"
Status: Recruiting | Type: Observational
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Collaborators: Prof. Otto Beisheim Foundation (Other)
Responsible Party: Principal Investigator, Ellen Greimel, Working group leader, LMU Klinikum
Other Study IDs: 24-0201 KB
Record Dates: First submitted 2024-09-27; First posted 2024-10-31 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Depressive Disorder; Depression; Depression in Children; Depression in Adolescence
Keywords: depression; prevention; web-based; adolescents; depression literacy; user experience; acceptance
MeSH Terms: conditions — Depressive Disorder; Depression

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: "ich bin alles" — The web-based information platform "ich bin alles" (www-ich-bin-alles.de) on depression and mental health in childhood and adolescence was developed by the Department of Child and Adolescent Psychiatry, Psychosomatics and Psychotherapy of the LMU Munich Hospital together with the Prof. Otto Beisheim Foundation. It is aimed at children and adolescents with depression, healthy children and adolescents and parents. The project focuses on education, prevention, support and destigmatisation through the transfer of evidence-based knowledge.

SUMMARY:
Using a multi-method approach, the aim of this study is to investigate the naturalistic user experience and acceptance of the German website "ich bin alles". This website offers evidence-based information about the symptoms, causes, course, treatment, and prevention of youth depression. Another aim of this study is to determine whether the desired target groups of the website can be reached.

DETAILED DESCRIPTION:
Depressive disorders are among the most common mental illnesses in children and adolescents and were already on the rise before the COVID-19 pandemic. This trend has been further exacerbated by the pandemic. Depression in adolescents is associated with particularly serious consequences, such as school and social problems, increased risk of suicide and impaired mental health in adulthood. If depression persists, the risk of chronification increases and continuous school attendance or continuation of vocational training is more difficult. The longer a depressive illness is not (effectively) treated, the lower the likelihood of remission and the higher the risk of chronification with further depressive episodes over the course of the illness. Although there are effective forms of treatment, in Germany only around 12% of adolescents with increased symptoms of depression seek professional treatment. The main barriers for adolescents to seek professional help include, for example, individual factors (low knowledge of mental disorders), social factors (e.g., perceived social stigmatisation) and systemic and structural barriers (e.g., limited access to professional help). In order to meet the need for action in a timely manner that meets the needs of the target group, the Department of Child and Adolescent Psychiatry of the Hospital of the LMU Munich and the Beisheim Foundation launched the innovative digital information portal "ich bin alles" ("I am everything"; www.ich-bin-alles.de) on depression and mental health in youth in 2021. Due to a sharp increase in online health information in recent years, the quality of this information and information portals has increasingly become the centre of attention. A review of the quality of mental health information websites found that many of the websites had shortcomings in terms of transparency, presentation and accuracy of content. These limitations were confirmed in a more recent study of depression websites. The comprehensibility of the content is also often limited, especially for users with a lower level of education and/or health literacy.

Due to the high relevance of comprehensively evaluating web-based information services on mental health and mental illness, the aim of this study is to use established methods to learn more about the visitors of "ich bin alles" and their user experience. This study will build on the approach of previous studies on website evaluation, which usually follow a multi-method approach: The evaluation of website analyses using tools such as Matomo; as well as an online questionnaire. The study is intended to provide clues as to whether the "ich bin alles" information platform is a useful and trustworthy source of information for the target groups. The information obtained is of central importance for potential adaptations and optimizations of the "ich bin alles" website. Another aim of this study is to determine whether "ich bin alles" can actually reach its desired target groups. The results of the data collection also provide an important basis for future approaches aimed at informing children, young people and their parents about mental health issues and mental illness in a way that is appropriate for the target group.

ELIGIBILITY:
Inclusion Criteria:

* 40 seconds website-use

Exclusion Criteria:

* no exclusion criteria

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: users of the website "ich bin alles"
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-06-20 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
The characteristics of the people who are interested in "ich bin alles" (i.e. the users) - Assessed via self-designed questionnaire | post (40 seconds after Website-use)
Perception of the users of website content - Assessed via WEB-CLIC-S | post (40 seconds after Website-use)
Perceived Website Usability - Assessed via Perceived Website Usability - German | post (40 seconds after Website-use)
Visual Aesthetics of Website - Assessed via Visual Aesthetics of Website Inventory - Short | post (40 seconds after Website-use)
Overall impression - assessed via a single item (school grade) | post (40 seconds after Website-use)
Intentions to act - Assessed via Scale assessing the intention to revisit the website | post (40 seconds after Website-use)

SECONDARY OUTCOMES:
specific data collected for "ich bin alles" with Matomo | 45 months (from launch of the website until anticipated study completion)
  Title of the pages accessed (page title)
specific data collected for "ich bin alles" with Matomo | 45 months (from launch of the website until anticipated study completion)
  Location of the users: Country, region, city, approximate latitude and longitude (geolocation)
specific data collected for "ich bin alles" with Matomo | 45 months (from launch of the website until anticipated study completion)
  Number of the website users
specific data collected for "ich bin alles" with Matomo | 45 months (from launch of the website until anticipated study completion)
  How the users accessed the website (e.g. Google search or Social Media link)
specific data collected for "ich bin alles" with Matomo | 45 months (from launch of the website until anticipated study completion)
  How much time the users spend on the website

CONTACTS AND LOCATIONS:
Overall Officials: Gerd Schulte-Körne, Prof. Dr., Study Director — Department of Child and Adolescent Psychiatry, Psychosomatics and Psychotherapy, LMU University Hospital
Locations (1):
- LMU University Hospital, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.ich-bin-alles.de/